CLINICAL TRIAL: NCT01277666
Title: A Randomised, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy and Safety of GSK1605786A in the Treatment of Subjects With Moderately-to-Severely Active Crohn's Disease
Brief Title: A Study to Investigate the Efficacy and Safety of GSK1605786A in the Treatment of Subjects With Moderately-to-Severely Active Crohn's Disease
Acronym: SHIELD-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114151
Record Dates: First submitted 2011-01-13; First posted 2011-01-17 (Estimated); Results first posted 2017-09-19 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-07

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; capsule; GSK1605786A; quality of life; inflammatory bowel disease; oral therapy
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — CCX282-B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): orally administered
  Interventions: Drug: Placebo
- GSK1605786A 500mg once daily (Experimental): orally administered
  Interventions: Drug: GSK1605786A
- GSK1605786A 500mg twice daily (Experimental): orally administered
  Interventions: Drug: GSK1605786A

INTERVENTIONS:
Drug: GSK1605786A — 500 mg twice daily, administered orally for 12 weeks
  Arms: GSK1605786A 500mg twice daily
Drug: GSK1605786A — 500 mg once daily, administered orally for 12 weeks
  Arms: GSK1605786A 500mg once daily
Drug: Placebo — Placebo capsules, administered orally for 12 weeks
  Arms: Placebo

SUMMARY:
This is a randomised, double-blind, placebo-controlled study to evaluate the efficacy and safety of two doses (500 mg once daily and 500 mg twice daily) of GSK1605786A as compared to placebo over 12 weeks in adult subjects with moderately-to-severely active Crohn's disease. Efficacy will be assessed by proportion of subjects achieving response, defined as a decrease in Crohn's Disease Activity Index (CDAI) score of at least 100 points (clinical response). Clinical remission (CDAI score less than 150 points) will be evaluated as a key secondary endpoint. Safety will be assessed by recording of adverse events, clinical laboratory parameters, vital signs and electrocardiogram (ECG). Population pharmacokinetics will evaluate the two doses of GSK1605786A. Health outcomes assessments will include changes in Inflammatory Bowel Disease Questionnaire (IBDQ), Short Form-36 version 2 (SF-36v2), EQ-5D and Work Productivity and Activity Impairment-CD (WPAI-CD) and receipt of disability.

DETAILED DESCRIPTION:
This is a multi-centre, randomised, double-blind, placebo-controlled, parallel group study to evaluate the efficacy of two oral doses of GSK1605786A (500 mg once daily, 500 mg twice daily) as compared to placebo in the induction of clinical response over a 12-week treatment period in subjects with moderately-to-severely active Crohn's disease. Secondary objectives will include assessment of the safety and evaluation of the efficacy in induction of remission.

The study is planned to randomise approximately 600 subjects (200 subjects/group) with active Crohn's disease, diagnosed for at least 4 months with a documented history of disease in the small and/or large intestine, and characterised by a Crohn's Disease Activity Index (CDAI) score between 220 to and 450, inclusive. Subjects must have reported an inadequate response or intolerance to Crohn's disease treatment with corticosteroids or immunosuppressants. Inclusion of subjects who received prior treatment with a biologic anti-tumour necrosis factor (TNF) agent will be limited to approximately 50% of the study population. All subjects are required to have a diagnosis with identification of anatomic location of Crohn's disease, which has been established by visualisation of the gastrointestinal tract within 12 months of screening. Subjects who have not had a visualisation of the gastrointestinal tract within 12 months are required to undergo an endoscopic assessment during the screening period. Subjects will be required to have evidence of current active inflammation at the time of randomisation either by endoscopy or by inflammatory biomarkers [elevated C-reactive protein (CRP) greater than the upper limit of normal (ULN) plus a positive faecal calprotectin test]. Subjects who do not meet the requirements based on inflammatory biomarker test results will be required to qualify based on endoscopic assessment during screening. Subjects will be allowed to participate in the study while continuing on stable doses of agents typically used to treat Crohn's disease. Following the screening period, subjects will be randomised at baseline to receive blinded treatment with one of two doses of GSK1605786A (500 mg once daily or twice daily) or placebo for 12 weeks. Response and remission endpoints, using the CDAI, will be evaluated at Weeks 4, 8 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 years or older
* Written informed consent
* Diagnosis of Crohn's disease for greater than 4 months duration with small bowel and/or colonic involvement
* Confirmation of Crohn's disease established by visualisation of the gastrointestinal tract within the 12 months prior to screening or by screening endoscopy at study entry
* History of inadequate response and/or intolerance/adverse event leading to discontinuation of either corticosteroids or immunosuppressants
* Moderately-to-severely active disease characterised by a CDAI score between 220 and 450, inclusive, at Baseline
* Confirmation of current active Crohn's disease by screening endoscopy or inflammatory biomarkers [elevated C-reactive protein (greater than upper limit of normal) plus positive test for faecal calprotectin] at Screening
* Stable doses of permitted concomitant medications or having previously received, but are not currently receiving, medications for Crohn's disease
* Demonstrated ability to comply with Crohn's disease symptom recording using the interactive voice response system
* Females of child-bearing potential must be sexually inactive or commit to consistent and correct use of a contraceptive method of birth control with a failure rate of less than 1% for the duration of this study

Exclusion Criteria:

* If female: pregnant, has a positive pregnancy test or is breast-feeding
* Diagnosis of coeliac disease, follow a gluten-free diet to manage symptoms, or positive test for coeliac disease
* Diagnosis of ulcerative or indeterminate colitis
* Enterocutaneous, abdominal or pelvic fistulae with abscesses or fistulae likely to require surgery during the study period
* Bowel surgery, other than appendectomy, within 12 weeks prior to screen and/or has surgery planned or deemed likely for Crohn's disease during the study period
* Extensive colonic resection, subtotal or total colectomy
* Presence of ileostomies, colostomies or rectal pouches
* Known fixed symptomatic stenoses
* History of more than 3 small bowel resections or diagnosis of short bowel syndrome
* Chronic use of narcotics for chronic pain defined as daily use of one or more doses of narcotic containing medication
* Use of prohibited medications, including enteral feeding or elemental diet, within their specified time frames

  1. Biologic use: Use of any biologic (tumour necrosis factor inhibitor or natalizumab) within 8 weeks prior to screening
  2. Corticosteroid use: Use of parenteral glucocorticoids within 4 weeks prior to screening
  3. Immunospressant use: Use of cyclosporine, tacrolimus, sirolimus or mycophenolate mofetil within 4 weeks prior to screening
  4. Intravenous antibiotic use: Use of intravenous antibiotics for Crohn's disease within 4 weeks prior to screening
  5. Use of rectal treatment with 5-ASA or corticosteroid enemas/suppositories within 2 weeks prior to screening
  6. Use of tube or enteral feeding, elemental diet, or parenteral alimentation within 2 weeks prior to screening
  7. Leukocytapheresis or granulocytapheresis within 2 weeks prior to screening
* Positive immunoassay for Clostridium difficile
* Known human immunodeficiency virus (HIV) infection
* Known varicella, herpes zoster, or other severe viral infection within 6 weeks of screening
* Immunisation with a live vaccine within 4 weeks of screening, with the exception of influenza vaccine
* Active or latent tuberculosis infection
* Current sepsis or infections requiring intravenous antibiotic therapy for more than 2 weeks
* Evidence of hepatic dysfunction, viral hepatitis, or current or chronic history of liver disease including non-alcoholic steatohepatitis (NASH)
* Positive test for Hepatitis B or Hepatitis C antibody at screening
* Corrected QT interval of ECG (electrocardiogram) greater than or equal to 450 milliseconds
* Concurrent illness or disability that may affect the interpretation of clinical data, or otherwise contraindicates participation in this clinical study
* History or evidence of adenomatous colonic polyps that have not been removed
* History of evidence of colonic mucosal dysplasia
* Current evidence of, or has been treated for a malignancy within the past five years (other than localised basal cell, squamous cell skin cancer, cervical dysplasia, or any cancer in situ that has been resected)
* Any previous participation in a clinical study of GSK1605786A (formerly ChemoCentryx compound CCX282-B)
* Medical history of sensitivity to any of the components of GSK1605786A
* Use of any investigational product within 30 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2010-12-20 (Actual); Primary Completion 2013-07-11 (Actual); Study Completion 2013-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (189):
- United States (46):
  - GSK Investigational Site, Little Rock, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Lakewood, Colorado
  - GSK Investigational Site, Littleton, Colorado
  - GSK Investigational Site, Hamden, Connecticut
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Maitland, Florida
  - GSK Investigational Site, Port Orange, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Oak Lawn, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Hammond, Louisiana
  - GSK Investigational Site, Monroe, Louisiana
  - GSK Investigational Site, Chevy Chase, Maryland
  - GSK Investigational Site, Towson, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Chesterfield, Michigan
  - GSK Investigational Site, Troy, Michigan
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Tupelo, Mississippi
  - GSK Investigational Site, Lee's Summit, Missouri
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Egg Harbor City, New Jersey
  - GSK Investigational Site, Voorhees Township, New Jersey
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Pasadena, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Seattle, Washington
- Australia (7):
  - GSK Investigational Site, Bankstown, New South Wales
  - GSK Investigational Site, Hersten, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Kurralta Park, South Australia
  - GSK Investigational Site, Fitzroy, Victoria
  - GSK Investigational Site, Prahran, Victoria
  - GSK Investigational Site, Fremantle, Western Australia
- Austria (3):
  - GSK Investigational Site, Hall in Tirol
  - GSK Investigational Site, Linz
  - GSK Investigational Site, Vienna
- Belgium (7):
  - GSK Investigational Site, Bonheiden
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Kortrijk
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Roeselare
- Canada (16):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Abbotsford, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Richmond Hill, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Lévis, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
- Czechia (5):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Ostrava - Vitkovice
  - GSK Investigational Site, Prague
- Denmark (5):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Aarhus
  - GSK Investigational Site, Herlev
  - GSK Investigational Site, Hvidovre
  - GSK Investigational Site, Odense
- France (9):
  - GSK Investigational Site, Amiens
  - GSK Investigational Site, Clichy
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Saint-Priest-en-Jarez
  - GSK Investigational Site, Vandœuvre-lès-Nancy
- Germany (15):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Braunschweig, Lower Saxony
  - GSK Investigational Site, Brinkum/Stuhr, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Minden, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Ludwigshafen am Rhein, Rhineland-Palatinate
  - GSK Investigational Site, Dessau, Saxony-Anhalt
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Jena, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Hungary (3):
  - GSK Investigational Site, Békéscsaba
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Szekszárd
- Israel (6):
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Holon
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Tel Aviv
- Italy (4):
  - GSK Investigational Site, Palermo, Sicily
  - GSK Investigational Site, Genova
  - GSK Investigational Site, Modena
  - GSK Investigational Site, Roma
- Japan (9):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- Netherlands (5):
  - GSK Investigational Site, Almere Stad
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Ede
  - GSK Investigational Site, Heerlen
  - GSK Investigational Site, Rotterdam
- New Zealand (6):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Dunedin
  - GSK Investigational Site, Hamilton
  - GSK Investigational Site, Lower Hutt
  - GSK Investigational Site, Otahuhu
  - GSK Investigational Site, Tauranga
- Norway (6):
  - GSK Investigational Site, Ålesund
  - GSK Investigational Site, Bodø
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Tromsø
  - GSK Investigational Site, Trondheim
  - GSK Investigational Site, Tønsberg
- Poland (6):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Sopot
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Wroclaw
- Slovakia (5):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Nitra
  - GSK Investigational Site, Nové Mesto nad Váhom
  - GSK Investigational Site, Prešov
  - GSK Investigational Site, Trnava
- South Africa (4):
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Claremont
  - GSK Investigational Site, Observatory
  - GSK Investigational Site, Parktown
- South Korea (4):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Wŏnju
- Spain (5):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Elche
  - GSK Investigational Site, Galdakao/Vizcaya
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Sabadell (Barcelona)
- Sweden (4):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Umeå
- United Kingdom (9):
  - GSK Investigational Site, Harrow, Middlesex
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Nottingham
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Salford

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 608 participants with moderately-to-severely active Crohn's disease were enrolled in this study. The study was conducted at 162 centres in 23 countries, with sites in North America, Europe, Israel, South Africa, Japan, Australia, Korea and New Zealand. Study duration was from 20 December 2010 to 11 July 2013.
Pre-assignment Details: Of the total 1205 participants screened, 597 were screen failures and 608 participants were randomized in the study.
Groups:
- Placebo: Eligible participants were randomized at baseline (Week 0) to receive matching placebo orally for 12 weeks treatment period
- GSK1605786A 500 mg Once Daily: Eligible participants were randomized at baseline (Week 0) to receive GSK1605786A 500 milligram (mg) once daily hard gelatin capsules orally for 12 weeks treatment period
- GSK1605786A 500 mg Twice Daily: Eligible participants were randomized at baseline (Week 0) to receive GSK1605786A 500 mg twice daily hard gelatin capsules orally for 12 weeks treatment period
Period: Overall Study
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg Twice Daily
Started | 203 | 203 | 202
Completed | 158 | 144 | 153
Not Completed | 45 | 59 | 49
Not completed — Adverse Event | 26 | 25 | 20
Not completed — Lack of Efficacy | 8 | 20 | 12
Not completed — Protocol Violation | 2 | 3 | 2
Not completed — Protocol Defined Stopping criteria | 1 | 2 | 6
Not completed — Lost to Follow-up | 1 | 1 | 2
Not completed — Withdrawal by Subject | 7 | 8 | 6
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- GSK1605786A 500 mg Once Daily: Eligible participants were randomized at baseline (Week 0) to receive GSK1605786A 500 mg once daily hard gelatin capsules orally for 12 weeks treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg Twice Daily | Total
Number analyzed (Participants) | 203 | 203 | 202 | 608
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.1 (12.62) | 37.0 (12.60) | 35.9 (12.51) | 36.3 (12.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 130 | 106 | 339
  Male | 100 | 73 | 96 | 269
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 3
  Asian | 18 | 21 | 17 | 56
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 4 | 2 | 13
  White | 177 | 177 | 179 | 533
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Crohn's Disease Activity Index (CDAI) Response at Week 12
Description: CDAI is a number which consists of information collected from a 7-day diary from the participants regarding symptoms. Remission is considered a score of 150 or less. Active disease is considered 200 or greater. A response to therapy is considered a decline in CDAI score of 70-points from baseline. The score was algorithmically derived from the sum of participant reported Crohn's disease symptoms recorded over 7 days and investigator recorded assessments of the participant's condition, laboratory parameters and use of anti-diarrhoeal medication. CDAI score was calculated based on the data collected in the diary card. The total CDAI score ranged from 0 to approximately 600, where higher scores indicate more severe disease. Both participants and investigators made their entries via IVRS each evening before going to bed. Percentage of participants with CDAI response at Week 12 was presented.
Time Frame: Week 12
Population: The intent to treat population comprised of all participants randomized to double-blind treatment for 12 weeks.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg Twice Daily
Number analyzed (Participants) | 203 | 203 | 202
Percentage of participants | 25.1 [19.2 to 31.1] | 27.6 [21.4 to 33.7] | 27.2 [21.1 to 33.4]
Statistical Analysis 1: Comparison: Placebo vs GSK1605786A 500 mg Once Daily; comparison of Placebo and GSK1605786A 500 mg once daily; Test type: Superiority or Other; p = 0.546, Mantel Haenszel; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [-6.1 to 11.0]
Statistical Analysis 2: Comparison: Placebo vs GSK1605786A 500 mg Twice Daily; comparison of Placebo and GSK1605786A 500 mg twice daily; Test type: Superiority or Other; p = 0.648, Mantel Haenszel; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [-6.5 to 10.7]

2. Secondary Outcome: Percentage of Participants With CDAI Remission at Week 12
Description: CDAI is a recognized scoring system to categorize disease severity with scores of >= 220 to <= 450 describing the moderately-to-severely active population. Clinical remission is defined as a CDAI score < 150 points if baseline CDAI is >= 150. If baseline CDAI is <150, the participant was not considered in remission. Participants with missing CDAI scores were considered not in remission according to the missing=no effect imputation. Percentage of participants in clinical remission at Week 12 was presented.
Time Frame: Week 12
Population: Intent to treat population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg Twice Daily
Number analyzed (Participants) | 203 | 203 | 202
Percentage of participants | 15.3 [10.3 to 20.2] | 13.3 [8.6 to 18.0] | 12.9 [8.3 to 17.5]
Statistical Analysis 1: Comparison: Placebo vs GSK1605786A 500 mg Once Daily; Test type: Superiority or Other; p = 0.592, Mantel Haenszel; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-8.8 to 4.8]
Statistical Analysis 2: Comparison: Placebo vs GSK1605786A 500 mg Twice Daily; Test type: Superiority or Other; p = 0.475, Mantel Haenszel; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-9.2 to 4.4]

3. Secondary Outcome: Percentage of Participants With a Clinical Response (CDAI Decrease From Baseline of >= 100 Points) at Both Week 8 and Week 12
Description: Responders were defined as participants with CDAI decrease from baseline of >= 100 points. CDAI is a recognized scoring system to categorize disease severity with scores of >= 220 to <= 450 describing the moderately-to-severely active population. The score was algorithmically derived from the sum of participant reported Crohn's disease symptoms recorded over 7 days and investigator recorded assessments of the participant's condition, laboratory parameters and use of anti-diarrhoeal medication. Both participants and investigators made their entries via IVRS each evening before going to bed. Percentage of participants with CDAI decrease from baseline of >=100 points was presented.
Time Frame: At Week 8 and 12
Population: Intent to treat population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg Twice Daily
Number analyzed (Participants) | 203 | 203 | 202
Percentage of participants | 15.8 [10.8 to 20.8] | 18.7 [13.4 to 24.1] | 19.3 [13.9 to 24.8]
Statistical Analysis 1: Comparison: Placebo vs GSK1605786A 500 mg Once Daily; Test type: Superiority or Other; p = 0.415, Mantel Haenszel; Mean Difference (Final Values) = 3.0, 95% CI 2-sided [-4.4 to 10.3]
Statistical Analysis 2: Comparison: Placebo vs GSK1605786A 500 mg Twice Daily; Test type: Superiority or Other; p = 0.354, Mantel Haenszel; Mean Difference (Final Values) = 3.5, 95% CI 2-sided [-3.9 to 10.9]

4. Secondary Outcome: Percentage of Participants Achieving Clinical Remission (CDAI <150 Points) at Both Week 8 and Week 12
Description: Clinical remission is defined as a CDAI score < 150 points if baseline CDAI is >= 150. If baseline CDAI is <150, the participant was not considered in remission. participants with missing CDAI scores were considered not in remission according to the missing=no effect imputation. Percentage of participants in clinical remission defined as a CDAI score of less than 150 points at other time points was presented.
Time Frame: Week 8 and 12
Population: Intent to treat population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg Twice Daily
Number analyzed (Participants) | 203 | 203 | 202
Percentage of participants | 7.9 [4.2 to 11.6] | 7.9 [4.2 to 11.6] | 6.9 [3.4 to 10.4]
Statistical Analysis 1: Comparison: Placebo vs GSK1605786A 500 mg Once Daily; Test type: Superiority or Other; p = 0.985, Mantel Haenszel; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-5.2 to 5.2]
Statistical Analysis 2: Comparison: Placebo vs GSK1605786A 500 mg Twice Daily; Test type: Superiority or Other; p = 0.709, Mantel Haenszel; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-6.1 to 4.1]

5. Secondary Outcome: Percentage of Participants With a Clinical Response (CDAI Decrease From Baseline of >=100 Points) at Week 8
Description: CDAI is a recognized scoring system to categorize disease severity with scores of >= 220 to <= 450 describing the moderately-to-severely active population. The score was algorithmically derived from the sum of participant reported Crohn's disease symptoms recorded over 7 days and investigator recorded assessments of the participant's condition, laboratory parameters and use of anti-diarrhoeal medication. Both participants and investigators made their entries via IVRS each evening before going to bed. Percentage of Participants with a clinical response CDAI decrease from baseline of >=100 points at Week 8 was presented.
Time Frame: Week 8
Population: Intent to treat population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg Twice Daily
Number analyzed (Participants) | 203 | 203 | 202
Percentage of Participants | 24.1 [18.3 to 30.0] | 26.1 [20.1 to 32.2] | 24.8 [18.8 to 30.7]
Statistical Analysis 1: Comparison: Placebo vs GSK1605786A 500 mg Once Daily; Test type: Superiority or Other; p = 0.633, Mantel Haenszel; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [-6.5 to 10.4]
Statistical Analysis 2: Comparison: Placebo vs GSK1605786A 500 mg Twice Daily; Test type: Superiority or Other; p = 0.889, Mantel Haenszel; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-7.8 to 9.0]

6. Secondary Outcome: Percentage of Participant Achieving Clinical Remission (CDAI <150 Points) at Week 8
Description: Clinical remission is defined as a CDAI score < 150 points if baseline CDAI is >= 150. If baseline CDAI is <150, the participant was not considered in remission. participants with missing CDAI scores were considered not in remission according to the missing=no effect imputation. Percentage of participants achieving clinical remission with CDAI <150 points at Week 8 was presented.
Time Frame: Week 8
Population: Intent to treat population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg Twice Daily
Number analyzed (Participants) | 203 | 203 | 202
Percentage of participants | 12.3 [7.8 to 16.8] | 10.3 [6.2 to 14.5] | 9.9 [5.8 to 14.0]
Statistical Analysis 1: Comparison: Placebo vs GSK1605786A 500 mg Once Daily; Test type: Superiority or Other; p = 0.541, Mantel Haenszel; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-8.1 to 4.2]
Statistical Analysis 2: Comparison: Placebo vs GSK1605786A 500 mg Twice Daily; Test type: Superiority or Other; p = 0.430, Mantel Haenszel; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-8.5 to 3.7]

7. Secondary Outcome: Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score at Both Weeks 8 and 12
Description: The IBDQ is a 32-item IBD-specific health related quality of life instrument evaluating general activities of daily living, intestinal function, social performance, personal interactions, and emotional status. Each item response was graded from 1 to 7 for each area evaluated. A higher score indicated better function in that area. Total IBDQ score was obtained by summing up scores for all 32 questions. Total IBDQ score ranged from 32 to 224. A higher score indicated better quality of life and lower score indicated worse quality of life. Day 1 assessment was considered as Baseline. Change from Baseline was calculated by subtracting value at Baseline from value at Weeks 8 and 12.
Time Frame: Baseline (Week 0), Week 8 and Week 12
Population: Intent to treat population. Only those participants available at specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg Twice Daily
Number analyzed (Participants) | 203 | 203 | 202
Score on scale
  Week 8: number analyzed (Participants) | 191 | 196 | 185
  Week 8 | 13.18 (1.728) | 12.06 (1.704) | 16.55 (1.757)
  Week 12: number analyzed (Participants) | 191 | 196 | 185
  Week 12 | 13.00 (1.889) | 12.66 (1.863) | 14.86 (1.921)
Statistical Analysis 1: Comparison: Placebo vs GSK1605786A 500 mg Once Daily; Week 8; Test type: Superiority or Other; p = 0.642, ANCOVA — P-values were obtained from an analysis of covariance model with baseline score as the covariate; Mean Difference (Net) = -1.13, 95% CI 2-sided [-5.89 to 3.64], Standard Error of Mean 2.426
Statistical Analysis 2: Comparison: Placebo vs GSK1605786A 500 mg Once Daily; Week 12; Test type: Superiority or Other; p = 0.898, ANCOVA — P-values were obtained from an analysis of covariance model with baseline score as the covariate; Mean Difference (Net) = -0.34, 95% CI 2-sided [-5.55 to 4.87], Standard Error of Mean 2.652
Statistical Analysis 3: Comparison: Placebo vs GSK1605786A 500 mg Twice Daily; Week 8; Test type: Superiority or Other; p = 0.173, ANCOVA — P-values were obtained from an analysis of covariance model with baseline score as the covariate; Mean Difference (Net) = 3.37, 95% CI 2-sided [-1.48 to 8.21], Standard Error of Mean 2.467
Statistical Analysis 4: Comparison: Placebo vs GSK1605786A 500 mg Twice Daily; Week 12; Test type: Superiority or Other; p = 0.493, ANCOVA — P-values were obtained from an analysis of covariance model with baseline score as the covariate; Mean Difference (Net) = 1.85, 95% CI 2-sided [-3.45 to 7.15], Standard Error of Mean 2.697

8. Secondary Outcome: Incidence of Adverse Events (AE) and Serious Adverse Events (SAE)
Description: Data for number of participants who presented one or more adverse events (serious or non serious) was reported. An AE was defined as any untoward medical occurrence (MO) in a participant temporally associated with the use of a medicinal product (MP), whether or not considered related to the MP and can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with its use. The SAE was any untoward MO that, at any dose, results in death, life threatening, persistent or significant disability/incapacity, results in or prolongs inpatient hospitalization, congenital abnormality or birth defect, that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition.
Time Frame: Up to Week 12
Population: The Safety population comprised of all participants in the intent to treat population except those who did not take at least one dose of investigational product.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg Twice Daily
Number analyzed (Participants) | 202 | 202 | 201
Participants
  AE | 141 | 148 | 157
  SAE | 18 | 12 | 12

ADVERSE EVENTS:
Time Frame: Up to Week 12
Description: Safety population was used to collects AEs
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg Twice Daily
All-Cause Mortality (participants affected / at risk) | 0/202 | 0/202 | 1/201
Serious Adverse Events (participants affected / at risk) | 18/202 | 12/202 | 12/201
Other Adverse Events (participants affected / at risk) | 77/202 | 82/202 | 100/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=202) | GSK1605786A 500 mg Once Daily (N=202) | GSK1605786A 500 mg Twice Daily (N=201)
Crohn's disease (Gastrointestinal disorders) | 5 | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal fistula (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 2
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Salmonellosis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Varicella (Infections and infestations) | 1 | 0 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Postoperative adhesion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 2
Body temperature increased (Investigations) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Prostatism (Reproductive system and breast disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Intermittent claudication (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=202) | GSK1605786A 500 mg Once Daily (N=202) | GSK1605786A 500 mg Twice Daily (N=201)
Headache (Nervous system disorders) | 31 (53) | 32 (53) | 28 (42)
Crohn's disease (Gastrointestinal disorders) | 20 (21) | 23 (27) | 18 (22)
Nasopharyngitis (Infections and infestations) | 18 (20) | 16 (18) | 20 (23)
Abdominal pain (Gastrointestinal disorders) | 13 (21) | 17 (19) | 23 (25)
Nausea (Gastrointestinal disorders) | 15 (15) | 19 (22) | 18 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (14) | 14 (17) | 10 (12)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 7 (10) | 23 (27)
Vomiting (Gastrointestinal disorders) | 4 (4) | 12 (14) | 15 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.